CLINICAL TRIAL: NCT00182936
Title: A Trial to Reduce Delirium in Aged Post Acute Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Paul B. Beeson Career Development Awards in Aging Research Program (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0040; AG17649
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-11-20 (Estimated); Status verified 2006-11

CONDITIONS: Delirium; Aging
Keywords: Cognition disorder; organic brain syndrome; patient care management; long term care; extended care facility
MeSH Terms: conditions — Delirium; Cognition Disorders

INTERVENTIONS:
Behavioral: Delirium Abatement Program

SUMMARY:
The purpose of this study is to develop a comprehensive Delirium Abatement Program of care of delirious patients in the post acute care setting and to evaluate its impact on persistence and severity of delirium and on functional recovery.

DETAILED DESCRIPTION:
Common, morbid, and costly, delirium affects one third of hospitalized elders, and plays a central role in the cascade of adverse events that leads to functional decline and loss of independence. Moreover, as acute care stays continue to shorten and evidence mounts that delirium may persist for many weeks, concern about delirium can no longer be confined to the hospital. It is believed that a Delirium Abatement Program may significantly reduce the persistence of delirium in post-acute settings, and thereby improve functional recovery both during the post-acute stay and after discharge.

The Delirium Abatement Program (DAP) will be designed to assist facility staff to 1) detect delirium among new admissions, 2) evaluate common underlying causes of delirium, 3) prevent complications commonly associated with delirium, and 4) restore delirious patients' cognitive, behavioral, social and self care functioning to baseline status.

This three year trial will enroll 500 delirious patients admitted to eight Boston area post-acute skilled nursing facilities. The DAP intervention will be carried out in four facilities. Four other facilities, matched to the intervention by demographic, facility, and clinical characteristics, will serve as controls. Patients will be recruited within 72 hours (maximum 120 hrs) of admission, assessed weekly while in the facility, and at one, three, and six months following admission.

ELIGIBILITY:
Inclusion Criteria:

* Admission to study site following acute care medical/surgical hospitalization
* Aged 65 or older
* English-speaking
* Communicative prior to acute illness
* Not admitted for terminal care (life expectancy greater than 6 months)
* Residence within 25 miles of research site

Exclusion Criteria:

* Significant hearing impairment which precludes interviews
* End stage dementia (complete ADL dependence)
* Previous study enrollment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500
Dates: Start 2000-05; Study Completion 2004-06

PRIMARY OUTCOMES:
Prevalence of delirium at two weeks after admission
Activities of Daily Living (ADL) functional improvement two weeks after admission
Full ADL functional recovery to pre-illness status three months after post-acute admission

SECONDARY OUTCOMES:
Examination of differences between patients in facilities receiving the Delirium Abatement Program and those not on additional outcomes of delirium persistence and ADL improvement one month following admission
Differences in delirium severity, length of post acute stay, and health care resource utilization

CONTACTS AND LOCATIONS:
Overall Officials: Edward Marcantonio, MD, SM, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Hebrew Rehabilitation Center for Aged, Boston, Massachusetts, United States

REFERENCES:
- [Background] Lipowski ZJ. Delirium in the elderly patient. N Engl J Med. 1989 Mar 2;320(9):578-82. doi: 10.1056/NEJM198903023200907. No abstract available. PMID 2644535
- [Background] Marcantonio ER, Flacker JM, Michaels M, Resnick NM. Delirium is independently associated with poor functional recovery after hip fracture. J Am Geriatr Soc. 2000 Jun;48(6):618-24. doi: 10.1111/j.1532-5415.2000.tb04718.x. PMID 10855596
- [Background] Levkoff SE, Evans DA, Liptzin B, Cleary PD, Lipsitz LA, Wetle TT, Reilly CH, Pilgrim DM, Schor J, Rowe J. Delirium. The occurrence and persistence of symptoms among elderly hospitalized patients. Arch Intern Med. 1992 Feb;152(2):334-40. doi: 10.1001/archinte.152.2.334. PMID 1739363
- [Result] Marcantonio ER, Simon SE, Bergmann MA, Jones RN, Murphy KM, Morris JN. Delirium symptoms in post-acute care: prevalent, persistent, and associated with poor functional recovery. J Am Geriatr Soc. 2003 Jan;51(1):4-9. doi: 10.1034/j.1601-5215.2002.51002.x. PMID 12534838
- [Result] Marcantonio ER, Kiely DK, Simon SE, John Orav E, Jones RN, Murphy KM, Bergmann MA. Outcomes of older people admitted to postacute facilities with delirium. J Am Geriatr Soc. 2005 Jun;53(6):963-9. doi: 10.1111/j.1532-5415.2005.53305.x. PMID 15935018
- [Result] Simon SE, Bergmann MA, Jones RN, Murphy KM, Orav EJ, Marcantonio ER. Reliability of a structured assessment for nonclinicians to detect delirium among new admissions to postacute care. J Am Med Dir Assoc. 2006 Sep;7(7):412-5. doi: 10.1016/j.jamda.2006.02.006. Epub 2006 May 30. PMID 16979083
- [Result] Bergmann MA, Murphy KM, Kiely DK, Jones RN, Marcantonio ER. A model for management of delirious postacute care patients. J Am Geriatr Soc. 2005 Oct;53(10):1817-25. doi: 10.1111/j.1532-5415.2005.53519.x. PMID 16181185
- [Derived] Marcantonio ER, Bergmann MA, Kiely DK, Orav EJ, Jones RN. Randomized trial of a delirium abatement program for postacute skilled nursing facilities. J Am Geriatr Soc. 2010 Jun;58(6):1019-26. doi: 10.1111/j.1532-5415.2010.02871.x. Epub 2010 May 7. PMID 20487083